CLINICAL TRIAL: NCT00756964
Title: Effect of Rasburicase on Acute Kidney Injury, Kidney Function, the Incidence of Renal Replacement Therapy and All-cause Mortality Following Cardiac Surgery.
Brief Title: Lowering Serum Uric Acid to Prevent Acute Kidney Injury
Acronym: RasbAKI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: WIRB 20081132
Record Dates: First submitted 2008-09-19; First posted 2008-09-22 (Estimated); Results first posted 2012-09-03 (Estimated); Last update posted 2012-09-03 (Estimated); Status verified 2012-08

CONDITIONS: Hyperuricemia
Keywords: cardiac surgery; hyperuricemia
MeSH Terms: conditions — Hyperuricemia | interventions — rasburicase; Excipients

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rasburicase (Active Comparator): patients receiving rasburicase to lower serum uric acid
  Interventions: Drug: Rasburicase
- Placebo (Placebo Comparator): patients will receive a placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rasburicase — Rasburicase (Dose: 7.5mg in 50ml of normal saline administered over 30 minutes) or identical placebo will be administered as an (dosage form)intravenous infusion preoperatively.
  Other Names: urate oxidase enzyme
  Arms: Rasburicase
Drug: Placebo — Placebo drug (color-coded to appear identical to study drug) administered as an (dosage form) intravenous infusion preoperatively.
  Other Names: inactive ingredient
  Arms: Placebo

SUMMARY:
Acute kidney injury is associated with a rise in serum uric acid during cardiovascular surgery and can cause poor blood flow to the kidneys making them vulnerable to kidney injury. We hypothesize that hyperuricemia, particularly if chronic and marked, is a risk factor for acute kidney injury. The preoperative lowering of serum uric acid will reduce the incidence of acute kidney injury following cardiovascular surgery.

DETAILED DESCRIPTION:
The study will be a prospective, double-blind, placebo-controlled, randomized, clinical trial, initiated and implemented conjointly by the Nephrology and Cardiovascular Surgery Departments at Shands Hospital at the University of Florida in Gainesville, FL. We propose to study whether lowering uric acid provides significant renal and cardiovascular protection in subjects undergoing cardiovascular surgery. Up to 30 patients presenting for elective or urgent cardiovascular surgery with uric acid level > 6.5 mg/dl and estimated glomerular filtration of 30 - 60 ml/min will be included in the study. Patients recruitment will continue until up to 30 patients have completed the study, taking into account expected patient loss due to withdrawal of consent, incomplete study and other reasons.

Patients will be randomized to a control group or rasburicase group. Rasburicase or identical placebo will be administered to each group after randomization. A selected number of patients may undergo additional testing for mechanistic (non-clinical) secondary endpoints.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older, and
2. Undergoing elective cardiothoracic surgery(s), alone or in combination with other procedures/surgery(s): thoracic aortic aneurysm, cardiac valves, coronary artery bypass grafting, abdominal thoracic aneurysm, other CV surgery, and
3. Preoperative serum uric acid > 6.5 mg/dL, and
4. Preoperative estimated glomerular filtration rate of >30ml/min/1.73m2 or higher, but less than 60ml/min/1.73m2

Exclusion Criteria:

1. Prior history of allergy/adverse reaction to Rasburicase
2. History of any organ transplant
3. Preoperative intra-aortic balloon pump (IABP)
4. Known glucose 6-phosphate dehydrogenase (G6PD) deficiency
5. Current use of natriuretic peptides

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2008-10; Primary Completion 2011-07 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: A. Ahsan Ejaz, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

REFERENCES:
- [Background] Ejaz AA, Mu W, Kang DH, Roncal C, Sautin YY, Henderson G, Tabah-Fisch I, Keller B, Beaver TM, Nakagawa T, Johnson RJ. Could uric acid have a role in acute renal failure? Clin J Am Soc Nephrol. 2007 Jan;2(1):16-21. doi: 10.2215/CJN.00350106. Epub 2006 Dec 6. PMID 17699382

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from the Cardiovascular Surgery clinics. Written consents were obtained from all patients.
Pre-assignment Details: A large number of patients were screened to achieve the final participant numbers.
Groups:
- Rasburicase Group: The drug rasburicase was used in this group.
- Placebo Group: This group received an identical placebo of rasburicase.
Period: Overall Study
Arm/Group | Rasburicase Group | Placebo Group
Started | 13 | 13
Completed | 13 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rasburicase Group | Placebo Group | Total
Number analyzed (Participants) | 13 | 13 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 13 | 26
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 9 | 9 | 18
Region of Enrollment [Number; unit: participants]
  United States | 13 | 13 | 26

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Acute Kidney Injury (AKI).
Description: Acute kidney injury will be defined as an increase in serum creatinine of 0.3mg/dL from baseline or a 50% increase in serum creatinine from baseline values within 48 hours after surgery.
Time Frame: Within 48 hours postoperatively
Population: As no similar study has been performed, a power analysis could not be performed. As such, we decided to do a pilot study with 26 subjects and to set criteria to maximize the likelihood of seeing an effect.
Measure: Number; unit: Participants
Groups:
- Rasburicase Group: The patients received the drug rasburicase 7.5mg in 50mL of normal saline over 30 minutes period
- Placebo Group: The patients which received a placebo identical to rasburicase.
Arm/Group | Rasburicase Group | Placebo Group
Number analyzed (Participants) | 13 | 13
Participants | 13 | 13

ADVERSE EVENTS:
Time Frame: No Adverse Events occurred during the 15 months when data was collected.
Arm/Group | Rasburicase Group | Placebo Group
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 0/13 | 0/13

LIMITATIONS AND CAVEATS:
The limitation of the pilot study is that it was not powered to provide definite answers, an inherent limitation attributed to the absence of similar studies.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No